CLINICAL TRIAL: NCT00867386
Title: Desensitization for Highly Sensitized Recipients of Pancreas Transplantation
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Xunrong Luo, Associate Professor in Medicine-Nephrology, Microbiology-Immunology and Surgery-Organ Transplantation, Northwestern University
Other Study IDs: STU 14940; CNV0058087 (Other: Office for Sponsored Research, Northwestern University)
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Type 1 Diabetes; Rejection of Pancreas Transplant; Desensitization
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study for patients with type 1 diabetes, whom are already scheduled to have desensitization treatment to help increase the chance of receiving a pancreas transplant.The study staff will be looking at medical records in order to collect past, present and future information for each subject's medical condition and/or transplant. There are no additional study tests, procedures or devices needed for our analysis.

DETAILED DESCRIPTION:
Please note that this study is observational. The treatment of each patient will be at the discretion of the care physician. The study investigators will ONLY be performing data collection and analysis.

Post transplant all patients will receive one additional cycle of plasma exchange with a moderate dose of Intravenous Immunoglobulin (IVIg) (0.4 mg/Kg). Antibody titers will be monitoring prior to plasma exchange and immediately following the treatment. At this point, since donor antigens are known, only antibodies to these antigens will be tested to minimize cost. We anticipate that in some patients, especially if the original titer of donor-specific antibody (DSA) was high (> 1:128), a rise in DSA will be observed following transplant. If indeed DSA will be present, additional monitoring will be initiated and the patient will be treated further with plasma exchange/IVIg cycles, with antibody monitoring before and immediately after each cycle. If no DSA are detected, patients will be monitoring on a every other day schedule for the first week; weekly for the next 3 weeks and monthly up to 6 months post transplant. Additional testing will be performed in the event of any clinical evidence of graft dysfunction, or following sever infection events.

Patient will be followed to 12 month post transplant or until one of the end points is reached:

1. pancreas graft failure: defined by return of hyperglycemia and resume of insulin therapy;
2. patient death due to all causes with functioning graft

ELIGIBILITY:
Inclusion Criteria:

* Pancreas transplant recipients with elevated panel reactive antibody levels of >50% and who have received desensitization treatment and subsequently receive their transplantation at Northwestern Memorial Hospital (NMH).

Exclusion Criteria:

* No Exclusion criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of type 1 diabetes who are highly sensitized (defined as having panel reactive antibody (PRA) level >50%) who underwent successful desensitization treatment followed by a deceased donor pancreas transplantation at NMH .
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-12; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Success of surgical engraftment. | Post-operative day 1
  This is measured by standard blood flow perfusion scan. Adequate blood flow is demonstrated by appropriate radioactive tracer uptake by the pancreas allograft. Lack of blood flow will prompt immediate surgical intervention.
Track the improvement of glycemic control. | Standard-of-care labs throughout duration of study
  Standard of care laboratory values measured routinely include: fasting and post-prandial glucose determination, serum C-peptide levels, improvement of Hemoglobin (A1C) levels post-transplant.
Rejection free graft survival. | 12 Month follow-up from baseline
  Serum amylase & lipase measured. Rising levels/aberrant glycemic control may indicate allograft rejection. Treatment - pancreas allograft rejection: 1) diagnosed by pancreas allograft biopsy; 2) if rejection, staining for C4d, repeat to DSA to determine rejection (acute antibody meditated humoral vs. acute cellular); 3) acute humoral rejection treated w/plasma exchange, then by Intravenous Immunoglobulin (IVIg) (0.5 gm/kg) every other day, daily polyclonal anti-thymocyte globulin (ATG) at 1.25 mg/kg. Treatment duration based on clinical response. Baseline immunosuppressive medications maintained during treatment.
Patient and graft survival. | At 12 Month follow-up
  Patient and graft survival will be calculated at this time.

SECONDARY OUTCOMES:
Tracking infection risks | Standard of care benchmarks through 12 months
  Screening for viral infections will be performed according to standard of care protocol. Asymptomatic or symptomatic Cytomegalovirus (CMV) viremia will be treated in consultation with Transplant Infectious Diseases Services. Testing for bacterial and fungal infections will be guided by clinical suspicion. Active infection will again be treated in consultation with the Transplant Infectious Diseases Service.
Bleeding complications | At 12 Months follow-up time points
  Though increased risks for bleeding have been associated with repeated plasma exchanges that deplete clotting factors, review to evaluate whether the limited number of plasma exchanges used in the standard of care protocols will show a minimal increase of risks for bleeding. At 12 Month follow-up time points, the number of bleeding episodes, their temporal relation to plasma exchange, and frequency of requirement for factor replacement will be analyzed.
Reversal or halting of diabetic complications | 0, 6, 12, 18, 24 Months
  For diabetic nephropathy, serum creatinine levels and urine microalbuminuria will be measured. the use of ACE inhibitors, angiotensin receptor blocker, or aldosterone receptor blocker will be noted. For diabetic retinopathy, patients will be referred to an ophthalmologist at the 12 and 24 Months time points to measure diabetic retinal changes based on the Early Treatment Diabetic Retinopathy Study (ETDRS) grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Xunrong Luo, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States